CLINICAL TRIAL: NCT05715047
Title: Reducing Persistent Fatigue Following Hematopoietic Stem Cell Transplantation
Brief Title: Intervention for Fatigue in HCT Recipients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Ashley M. Nelson, PhD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-513
Record Dates: First submitted 2023-01-27; First posted 2023-02-06 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Hematologic Cancer; Hematologic Malignancy
Keywords: Hematologic Cancer; Hematologic Malignancy; Hematopoietic Stem; HCT; Cognitive Behavioral Therapy; CBT
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT for Fatigue Program (Experimental): Screening for eligibility will use the Fatigue Symptoms Inventory (FSI) average severity item over the prior week. Scores of ≥4 of 0-10 will be invited to participate. 30 participants will be enrolled and will complete study procedures as outlined:
  * Baseline questionnaires.
  * 10 intervention sessions.
  * Questionnaires and surveys 3 and 5 months after enrollment.
  Interventions: Behavioral: CBT for Fatigue
- Usual Care (Active Comparator): Screening for eligibility will use the Fatigue Symptoms Inventory (FSI) average severity item over the prior week. Scores of ≥4 of 0-10 will be invited to participate. 30 participants will be enrolled and will complete study procedures as outlined:
  * Baseline questionnaires.
  * Receive adapted material from the MGH Bone Marrow Transplant Survivorship program outlining common contributors to fatigue after transplant and recommendations for management.
  * Questionnaires and surveys 3 and 5 months after enrollment.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: CBT for Fatigue — 10, individualized counseling sessions with a behavioral health counselor via Zoom platform.
  Arms: CBT for Fatigue Program
Behavioral: Usual Care — Standard transplant care.
  Arms: Usual Care

SUMMARY:
The purpose of this study is to assess whether a cognitive-behavioral therapy (CBT) for fatigue intervention is acceptable, feasible, and effective at managing fatigue and improving quality of life for patients following hematopoietic stem cell transplant (HCT).

DETAILED DESCRIPTION:
This research is being done to determine whether a cognitive-behavioral therapy (CBT) for fatigue intervention is feasible and effective at managing fatigue and improving quality of life in patients following hematopoietic stem cell transplant.

An open pilot of 6 participants will precede the randomized controlled trial. Study procedures for the open pilot include screening for eligibility, intervention Zoom sessions, questionnaires, and exit interviews with study staff.

Patients participating in the subsequent randomized controlled trial will be randomized into one of two study groups: CBT for fatigue intervention versus usual care.Study procedures include screening for eligibility, intervention Zoom sessions (intervention arm) or receipt of informational materials about fatigue (usual care arm), and completion of study questionnaires (after consent but before randomization and at approximately 3 and 5 months post-randomization).

This research study is expected to last about 3 years. It is expected about 66 people will take part in this research study.

The National Heart, Lung, and Blood Institute of the National Institute of Health is providing funding for this project.

ELIGIBILITY:
Inclusion Criteria

* adult patients (≥ 18 years)
* have the ability to speak and read English
* have undergone autologous or allogeneic transplant > 6 months prior to enrollment
* no evidence of disease relapse requiring therapy
* no new other malignancy requiring therapy after transplant
* report moderate to severe fatigue in the past week (FSI average severity item rating ≥ 4 of 0-10)
* are currently receiving their care at the MGH Blood and Marrow Transplant Clinic

Exclusion Criteria

* Patients with active cognitive impairment or uncontrolled psychiatric illness such as schizophrenia that the treating clinician believes prohibits informed consent or participation in the intervention
* Patients already receiving CBT care
* Patients living with untreated sleep apnea
* Patients with hypoxemia requiring oxygen supplementation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-11-29 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Rate of Satisfaction (Open Pilot only) | 3 month follow-up
  Acceptability is defined by at least 80% of participants reporting satisfaction on the Client Satisfaction Questionnaire (range 8-32, with higher scores representing higher satisfaction).
Rate of Enrollment | At recruitment
  The intervention will be deemed feasible if at least 60% of eligible participants are enrolled in the randomized trial.
Rate of Retention | Baseline (pre-randomization) up to 5 month follow-up
  The intervention will be deemed feasible if at least 70% of participants are retained in both arms of the randomized trial.
Rate of Intervention Completion | Baseline (pre-randomization) up to 3 month follow-up
  The intervention will be deemed feasible if at least 70% of participants enrolled complete at least 70% of intervention sessions of the randomized trial.

SECONDARY OUTCOMES:
Improvement of Fatigue | Baseline (pre-randomization) up to 5 month follow-up
  Fatigue will be assessed with the Functional Assessment of Chronic Illness Therapy-Fatigue subscale (FACIT-F). Longitudinal differences in fatigue will be investigated between study groups (FACIT-F score range 0-52, with lower scores indicating greater fatigue).
Improvement of Quality of Life | Baseline (pre-randomization) up to 5 month follow-up
  Quality of life will be assessed with the Functional Assessment of Cancer Therapy-Bone Marrow Transplant scale (FACT-BMT). Longitudinal differences in quality of life will be assessed between study groups (FACT-BMT score range 0-164, with higher scores indicating better quality of life).
Improvement of Mood | Baseline (pre-randomization) up to 5 month follow-up
  Improvement in anxiety and depression symptoms will be assessed with the PROMIS Anxiety and Depression Scales. Longitudinal differences in anxiety and depression symptoms will be assessed between study groups (PROMIS anxiety and depression scale scores range 8-40, with higher scores indicating worse anxiety and depression symptoms).

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Nelson, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation